CLINICAL TRIAL: NCT03594825
Title: Effect of Nighttime Valsartan on Prognosis of Nocturnal Hypertension Patients Undergoing Maintenance Hemodialysis
Brief Title: Nighttime Valsartan in Hemodialysis Hypertension
Acronym: NVHH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Cheng Wang, Director of Nephrology, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Valsartan
Record Dates: First submitted 2018-07-04; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Hypertension;Nephropathy
Keywords: Nocturnal Hypertension; Hemodialysis; Valsartan
MeSH Terms: conditions — Hypertensive Nephropathy | interventions — Valsartan; lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nighttime group (Experimental): patients with nocturnal hypertension taking valsartan at nighttime
  Interventions: Drug: Valsartan
- daytime group (Active Comparator): patients with nocturnal hypertension taking valsartan at daytime
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Valsartan — Different time of taking medicine
  Other Names: Novartis

SUMMARY:
Hypertension is one of the most important independent risk factors for the prognosis of maintenance hemodialysis patients. The incidence rate is high and the control rate is low. Nocturnal hypertension has been paid more attention in recent years. Compared to daytime blood pressure, nocturnal blood pressure is an independent and efficient prognostic indicator of hypertensive deaths and cardiovascular events, but it's lack of evidence about its impact on prognosis in hemodialysis patients and the effective treatment program. Our previous cohort study suggests that the incidence of nocturnal hypertension in patients with chronic kidney disease is up to 71.22%, with a significant increase as the decline of renal function, and more severe target organ damage in patients with nocturnal hypertension: the decrease of glomerular filtration rate, left ventricular hypertrophy, and the increase of all cause death and cardiovascular death. Our small sample size study show that night time antihypertensive drugs can better control blood pressure and delay the development of left ventricular hypertrophy. These preliminary results suggest that nocturnal hypertension is closely related to the prognosis of chronic renal disease. Taking antihypertensive drugs at night is one of the options for controlling nocturnal hypertension. However, it is not clear whether taking antihypertensive drugs at night can improve the prognosis of maintenance hemodialysis patients with nocturnal hypertension. To this end, we collect maintenance hemodialysis patients with nocturnal hypertension, and propose a time selective use of valsartan to intervene in nocturnal hypertension. By comparing the differences in the effects of valsartan on the prognosis of maintenance hemodialysis patients during the day or night, to further clarify the role of nocturnal hypertension in the prognosis of maintenance hemodialysis patients, whether controlling nocturnal hypertension can improve the prognosis of maintenance hemodialysis patients. The completion of the study will optimize the prevention and treatment of hypertension in maintenance hemodialysis patients, and provide an evidence for precise prevention and treatment of hypertension in maintenance hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old and <75 years.
2. Diagnosed as CKD 5th stage in accordance with the kdigo guide 2012 (egfr < 15 ml/ (min 1.73m2)).
3. Accept 2-3 times a week, 4h regular hemodialysis for >3 months.
4. Ambulatory blood pressure monitoring indicates nighttime blood pressure systolic blood pressure(SBP) > 120mmHg and / or diastolic blood pressure(DBP) > 70mmHg.

Exclusion Criteria:

1. Stop hemodialysis longer than one month more than 2 times.
2. Night learning or work, irregular rest for a long time.
3. Overloading capacity, ultrafiltration volume of each treatment >7% dry weight.
4. Persistent atrial fibrillation.
5. Severe anemia and severe dystrophy.
6. Patients with postural hypotension or symptomatic hypotension.
7. Severe side effects or contraindications of valsartan treatment.
8. Treatment of corticosteroids or other hormones at present.
9. Unable to cooperate or unable to tolerate ambulatory blood pressure monitoring.
10. Ineffective ambulatory blood pressure data.
11. The clinical data were incomplete during the treatment period; end-point events occurred within 6 months or follow-up time was less than 6 months.
12. In the first 3 months before admission, there were obvious cardiovascular and cerebrovascular diseases such as coronary syndrome, myocardial infarction or stroke.
13. There were complications such as vascular disease, infection and bleeding within 1 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
all-cause death | 5 years
  death caused by all causes
cardiovascular death | 5 years
  death caused by cardiovascular events, such as myocardial infarction, arrhythmia and heart failure
cerebrovascular death | 5 years
  death caused by cerebral vascular events, such as stroke

SECONDARY OUTCOMES:
Cardio cerebral vascular events | 5 years
  cardiovascular and cerebrovascular events that require hospitalization and lead to death or non death, including myocardial infarction, heart failure, stroke, vascular reconstruction, peripheral vascular disease, and non-traumatic amputation

OTHER OUTCOMES:
cardiovascular structural abnormalities | 5 years
  changes of carotid artery intima-media thickness and left ventricular mass index

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Wang, Director, Principal Investigator — Nephrology Department, the Fifth Affiliated Hospital of Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] K/DOQI Workgroup. K/DOQI clinical practice guidelines for cardiovascular disease in dialysis patients. Am J Kidney Dis. 2005 Apr;45(4 Suppl 3):S1-153. No abstract available. PMID 15806502
- [Background] Heerspink HJ, Ninomiya T, Zoungas S, de Zeeuw D, Grobbee DE, Jardine MJ, Gallagher M, Roberts MA, Cass A, Neal B, Perkovic V. Effect of lowering blood pressure on cardiovascular events and mortality in patients on dialysis: a systematic review and meta-analysis of randomised controlled trials. Lancet. 2009 Mar 21;373(9668):1009-15. doi: 10.1016/S0140-6736(09)60212-9. Epub 2009 Feb 25. PMID 19249092
- [Background] Agarwal R, Sinha AD. Cardiovascular protection with antihypertensive drugs in dialysis patients: systematic review and meta-analysis. Hypertension. 2009 May;53(5):860-6. doi: 10.1161/HYPERTENSIONAHA.108.128116. Epub 2009 Mar 9. PMID 19273737
- [Background] Nakai S, Masakane I, Akiba T, Iseki K, Watanabe Y, Itami N, Kimata N, Shigematsu T, Shinoda T, Syoji T, Syoji T, Suzuki K, Tsuchida K, Nakamoto H, Hamano T, Marubayashi S, Morita O, Morozumi K, Yamagata K, Yamashita A, Wakai K, Wada A, Tsubakihara Y. Overview of regular dialysis treatment in Japan (as of 31 December 2005). Ther Apher Dial. 2007 Dec;11(6):411-41. doi: 10.1111/j.1744-9987.2007.00523.x. PMID 18028170
- [Background] Agarwal R, Nissenson AR, Batlle D, Coyne DW, Trout JR, Warnock DG. Prevalence, treatment, and control of hypertension in chronic hemodialysis patients in the United States. Am J Med. 2003 Sep;115(4):291-7. doi: 10.1016/s0002-9343(03)00366-8. PMID 12967694
- [Background] Liu W, Ye H, Tang B, Song Z, Sun Z, Wen P, Yang J. Profile of interdialytic ambulatory blood pressure in a cohort of Chinese patients. J Hum Hypertens. 2014 Nov;28(11):677-83. doi: 10.1038/jhh.2014.41. Epub 2014 Jun 12. PMID 24919753
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force for the Management of Arterial Hypertension of the European Society of Hypertension and the European Society of Cardiology. 2013 ESH/ESC Practice Guidelines for the Management of Arterial Hypertension. Blood Press. 2014 Feb;23(1):3-16. doi: 10.3109/08037051.2014.868629. Epub 2013 Dec 20. No abstract available. PMID 24359485
- [Background] Hodgkinson J, Mant J, Martin U, Guo B, Hobbs FD, Deeks JJ, Heneghan C, Roberts N, McManus RJ. Relative effectiveness of clinic and home blood pressure monitoring compared with ambulatory blood pressure monitoring in diagnosis of hypertension: systematic review. BMJ. 2011 Jun 24;342:d3621. doi: 10.1136/bmj.d3621. PMID 21705406
- [Background] Fagard RH, Staessen JA, Thijs L. Relationships between changes in left ventricular mass and in clinic and ambulatory blood pressure in response to antihypertensive therapy. J Hypertens. 1997 Dec;15(12 Pt 1):1493-502. doi: 10.1097/00004872-199715120-00018. PMID 9431857
- [Background] Mancia G, Zanchetti A, Agabiti-Rosei E, Benemio G, De Cesaris R, Fogari R, Pessina A, Porcellati C, Rappelli A, Salvetti A, Trimarco B. Ambulatory blood pressure is superior to clinic blood pressure in predicting treatment-induced regression of left ventricular hypertrophy. SAMPLE Study Group. Study on Ambulatory Monitoring of Blood Pressure and Lisinopril Evaluation. Circulation. 1997 Mar 18;95(6):1464-70. doi: 10.1161/01.cir.95.6.1464. PMID 9118514
- [Background] Cuspidi C, Sala C, Valerio C, Negri F, Mancia G. Nocturnal blood pressure in untreated essential hypertensives. Blood Press. 2011 Dec;20(6):335-41. doi: 10.3109/08037051.2011.587280. Epub 2011 Jun 9. PMID 21651423
- [Background] Hoshide S, Ishikawa J, Eguchi K, Ojima T, Shimada K, Kario K. Masked nocturnal hypertension and target organ damage in hypertensives with well-controlled self-measured home blood pressure. Hypertens Res. 2007 Feb;30(2):143-9. doi: 10.1291/hypres.30.143. PMID 17460384
- [Background] Yano Y, Kario K. Nocturnal blood pressure and cardiovascular disease: a review of recent advances. Hypertens Res. 2012 Jul;35(7):695-701. doi: 10.1038/hr.2012.26. Epub 2012 Mar 1. PMID 22378470
- [Background] Clement DL, De Buyzere ML, De Bacquer DA, de Leeuw PW, Duprez DA, Fagard RH, Gheeraert PJ, Missault LH, Braun JJ, Six RO, Van Der Niepen P, O'Brien E; Office versus Ambulatory Pressure Study Investigators. Prognostic value of ambulatory blood-pressure recordings in patients with treated hypertension. N Engl J Med. 2003 Jun 12;348(24):2407-15. doi: 10.1056/NEJMoa022273. PMID 12802026
- [Background] Hansen TW, Li Y, Boggia J, Thijs L, Richart T, Staessen JA. Predictive role of the nighttime blood pressure. Hypertension. 2011 Jan;57(1):3-10. doi: 10.1161/HYPERTENSIONAHA.109.133900. Epub 2010 Nov 15. PMID 21079049
- [Background] Sarafidis PA, Persu A, Agarwal R, Burnier M, de Leeuw P, Ferro C, Halimi JM, Heine G, Jadoul M, Jarraya F, Kanbay M, Mallamaci F, Mark PB, Ortiz A, Parati G, Pontremoli R, Rossignol P, Ruilope L, Van der Niepen P, Vanholder R, Verharr MC, Wiecek A, Wuerzner G, London GM, Zoccali C. Hypertension in dialysis patients: a consensus document by the European Renal and Cardiovascular Medicine (EURECA-m) working group of the European Renal Association - European Dialysis and Transplant Association (ERA-EDTA) and the Hypertension and the Kidney working group of the European Society of Hypertension (ESH). J Hypertens. 2017 Apr;35(4):657-676. doi: 10.1097/HJH.0000000000001283. PMID 28157814
- [Background] Kishi T, Hirooka Y, Konno S, Sunagawa K. Angiotensin II receptor blockers improve endothelial dysfunction associated with sympathetic hyperactivity in metabolic syndrome. J Hypertens. 2012 Aug;30(8):1646-55. doi: 10.1097/HJH.0b013e328355860e. PMID 22728908
- [Background] Suzuki H, Kanno Y, Sugahara S, Ikeda N, Shoda J, Takenaka T, Inoue T, Araki R. Effect of angiotensin receptor blockers on cardiovascular events in patients undergoing hemodialysis: an open-label randomized controlled trial. Am J Kidney Dis. 2008 Sep;52(3):501-6. doi: 10.1053/j.ajkd.2008.04.031. Epub 2008 Jul 24. PMID 18653268
- [Background] Wang C, Zhang J, Liu X, Li CC, Ye ZC, Peng H, Chen Z, Lou T. Effect of valsartan with bedtime dosing on chronic kidney disease patients with nondipping blood pressure pattern. J Clin Hypertens (Greenwich). 2013 Jan;15(1):48-54. doi: 10.1111/jch.12021. Epub 2012 Oct 9. PMID 23282124